CLINICAL TRIAL: NCT00257517
Title: Home Surveillance and Feeding Strategies in Infants With Complex Single Ventricle
Brief Title: Multisite Feeding Study: Home Surveillance and Feeding Strategies in Infants With Complex Single Ventricle
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Martha L. Clabby, MD, Principal Investigator, Emory University
Other Study IDs: IRB00021873
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Congenital Disorders
Keywords: Congenital heart disease; Single ventricle; Infant feeding
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Heart Defects, Congenital; Univentricular Heart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will assess 75-100 patients for feeding issues following surgery for single ventricle.

DETAILED DESCRIPTION:
We wish to consent 75-100 subjects at Children's Healthcare of Atlanta.

If subjects take part in this study, the following will happen:

1. Prior to discharge, the parent/guardian will be given a home feeding log and
2. Parents will bring the feeding log to regularly scheduled clinic visits. Clinic staff will also weigh the child and measure head circumference at each clinic visit.
3. The investigators will look at the child's medical record to obtain other information including diagnosis, surgery, oxygen saturation levels and medications.
4. The parent/guardian will be asked to fill out a questionnaire about their stress and uncertainty caring for their baby after heart surgery. They will be asked to fill out the same questionnaire 3 times:

   * First time will be before they leave the hospital after the baby's surgery, while still a patient on the Cardiac Step Down Unit (CSU).
   * Second time will be at the Sibley Heart Center Cardiology clinic after they have been home for approximately 4 weeks.
   * Third time will be at the Sibley Heart Center Cardiology clinic after they have been home for approximately 12 weeks or at the time of the routine cardiac cath prior to their second stage surgery.

It should take about 15 minutes to fill out the questionnaire. The questionnaire is the only research procedure.

The data from the feeding log and clinic visits will be submitted to Cincinnati Children's, the primary site for this study.

ELIGIBILITY:
Inclusion Criteria:

* Single ventricle patients who have received the Norwood Stage I operation.

Exclusion Criteria:

* Infants with chromosomal anomalies or other non-cardiac conditions (cleft palate, necrotizing enterocolitis [NEC] or other gastrointestinal [GI] anomalies)
* Prematurity less than 37 weeks
* Infants greater than 30 days of age at Stage I palliation
* Parents who cannot read or understand questionnaires administered as a part of the study.

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: hypoplastic left heart syndrome
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-10; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
weight gain | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Martha Clabby, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States